CLINICAL TRIAL: NCT02004418
Title: A Prospective Single-Arm Phase I/II Study Using 11C-Choline PET Scans for Dose Escalated Hypofractionated Image Guided Inversely Planned Intensity Modulated External Beam Radiotherapy With Boost to PET Defined Dominant Intraprostatic Lesions and as a Predictive Factor for Biochemical Disease-Free Survival in Patients With Localized Prostate Cancer
Brief Title: A Study for Patients With Prostate Cancer to See Whether Delivering an Extra Dose of Radiation to Parts of the Body With More Cancer is Better Than Standard Treatment in Which the Same Dose of Radiation is Given Throughout the Prostate Gland
Acronym: PET PRO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-Amanie-02 (PET PRO)
Record Dates: First submitted 2013-11-15; First posted 2013-12-09 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Prostatic Neoplasms
Keywords: C-Choline PET scans; external beam radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will receive a fixed dose (400 MBq +/-10%) of 11C-Choline and PET/CT imaging with co-registration 3T MRI imaging prior to Enhanced EBRT and two further doses of 11C-Choline at two intervals (3 and 6 months) thereafter.
  Subjects with suitable intraprostatic lesion delineation with 11C-Choline will proceed to Enhanced EBRT, consisting of a dose prescription of 78 Gy in 25 fractions to the intraprostatic lesions and 68 Gy in 25 fractions (simultaneously) to the prostate gland. Subjects without suitable intraprostatic lesion delineation will be treated with Cross Cancer Institute standard of care EBRT and undergo follow-up for biochemical recurrence per protocol to determine the prognostic value of the baseline PET findings
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-Choline PET Scans (Experimental): Radioactive doses of 11C-Choline: 400 MBq ± 10% per injection, pre-radiation treatment and following treatment at 3 and 6 months
  Interventions: Radiation: 11C-Choline

INTERVENTIONS:
Radiation: 11C-Choline

SUMMARY:
Patients with localized prostate cancer are routinely treated with radiation therapy to the entire prostate gland. The investigators can identify where the cancer is concentrated in the prostate gland using a newer specialized imaging technique called 11C Choline PET (stands for choline positron emission tomography). This is different from the older type of PET scan that has been used in the past (called FDG PET) which has not been as accurate as the new PET scan for identifying where the cancer is in the prostate gland. It has also been shown that delivering higher doses of radiation to prostate cancer cells in the prostate have resulted in better cure rates in patients with prostate cancer. Therefore for goal number one the investigators want to give higher radiation dose to the prostate cancer cells. But the challenge has been that delivering higher doses of radiation to the prostate gland may also increase the chance of complications from the higher doses of radiation to the rectum, bladder and surrounding area. Therefore for goal number two the investigators want to minimize radiation dose to the rectum, bladder and surrounding area. 3-Tesla Magnetic Resonance Imaging (3T MRI) is a new kink of scan that will be used in this study to identify the urethra in the prostate so that the investigators can minimize the radiation dose to the urethra. The investigators believe the 3T MRI scan is able to point to the areas of cancer that may be able to predict how well the treatments may work, as well as which areas of the tumor appear to be responding to failing.

In this study, the investigators will keep the dose of radiation to the rectum and bladder as low as possible while increasing radiation dose to parts of the prostate with more cancer cells. The investigators will compare the cure rates in this study with the cure rates of other patients receiving the standard treatment in which the same dose of radiation is delivered throughout the prostate gland. The investigators will also compare the rates of complications in this study with the rates of complications in patients receiving the standard treatment in which the same dose of radiation is delivered throughout the prostate gland.

DETAILED DESCRIPTION:
This is a prospective, open label, non-randomized, single site, phase I/II study of the safety and utility of 11C-Choline PET scans for delineation of intraprostatic lesions in subjects with localized intermediate risk prostate cancer and subsequent Enhanced EBRT (External Beam Radiation Therapy) to monitor toxicity, therapeutic response and recurrence.

The estimated total number of subjects required for protocol enrollment and baseline 11C-Choline PET scans is 63; however, the protocol will complete accrual only when 29 subjects have commenced Enhanced EBRT or the outlined stopping rules require a halt to accrual. Twenty-nine (29) subjects treated with Enhanced EBRT are required to assess the toxicity of this treatment based on the statistical analysis outlined in the protocol. Subjects will receive a fixed dose (400 MBq, 10%) of 11C-Choline and PET/CT imaging with co-registration 3T MRI imaging prior to Enhanced EBRT and two further doses of 11C-Choline at two intervals (3 and 6 months) thereafter.

Subjects with suitable intraprostatic lesion delineation with 11C-Choline will proceed to Enhanced EBRT, consisting of a dose prescription of 78 Gy in 25 fractions to the intraprostatic lesions and 68 Gy in 25 fractions (simultaneously) to the prostate gland. Subjects without suitable intraprostatic lesion delineation will be treated with Cross Cancer Institute standard of care EBRT and undergo follow-up for biochemical recurrence per protocol to determine the prognostic value of the baseline PET findings.

Subjects will be monitored for 11C-Choline safety and efficacy and for EBRT safety / toxicity and efficacy.

11C-Choline PET image intraprostatic lesion(s) will be analyzed by the relative uptake scores (RUS), tumor to background ratios (T/B) and SUVmax parameters. Adequate delineation will be determined by a lesion with tumor to background ration ≥2. This is defined in section 10.

11C-Choline PET image parameters will be correlated with other measures of progression and survival including biochemical disease free survival as indicators of Enhanced EBRT response.

Efficacy of 11C-Choline delineated Enhanced EBRT will be evaluated by progression and survival analysis compared to historical data from this population.

Safety of 11C-Choline will be determined by: vital signs, blood hematology and clinical biochemistry profile (pre-injection, post-imaging) and adverse event collection.

Safety/toxicity of 11C-Choline delineated Enhanced EBRT will be determined by adverse event collection, primarily for genitourinary and gastrointestinal toxicity and compared to historical data from this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Biopsy proven prostate cancer with an intermediate risk feature defined as

   1. Gleason score 7, PSA <20, T1-T2C or
   2. Gleason score 6, PSA 10-20, T1-T2C or
   3. Gleason Score 6 or 7, PSA <20, T2C
3. Localized disease based on staging investigations including bone scan, CT abdomen and pelvis, and any other clinically indicated staging investigations
4. Eligible for curative intent external beam radiotherapy
5. Able and willing to follow instructions and comply with protocol
6. Provide written informed consent prior to participation in the study
7. Karnofsky Performance Scale Score 70-100

Exclusion Criteria:

1. Have had a 11C-Choline PET scan performed within 4 weeks after any biopsies of the prostate (due to concern that acute post biopsy intraprostatic changes may affect scan accuracy)
2. BMI ≥ 30
3. The presence of a hip prosthesis
4. Bilirubin ≥ 20 µmol/L
5. AST or ALT ≥ 5 times the upper limits of normal
6. Serious medical conditions which may prevent a patient from tolerating therapy such as: congestive heart failure, unstable angina, unstable ventricular arrhythmia, uncontrolled psychiatric conditions, serious infections and/or uncontrolled diabetes.
7. Metastatic disease
8. Prostate cancer with only low risk features or any high risk feature with a PSA ≥20 or T3 disease
9. A history of previous carcinoma except for basal cell carcinoma
10. Age < 18 years
11. Prior treatment with hormonal therapy
12. AUA prostate symptom score > 20
13. Crohn's disease or ulcerative colitis
14. Patient is unable to comply adequately iwth bowel or bladder prep during CT simulation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2019-11 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Determine the toxicity profile of 11C-Choline administration in PET scans, therapeutic response and biochemical recurrence in patients treated with EBRT. | After 3 months
Determine the toxicity profile of 11C-Choline administration in PET scans, therapeutic response and biochemical recurrence in patients treated with EBRT | After 3 years
Determine the toxicity profile of 11C-Choline administration in PET scans, therapeutic response and biochemical recurrence in patients treated with EBRT | After 5 years

SECONDARY OUTCOMES:
Intraprostatic lesion delineation capabilities of 11C-Choline in selected prostate cancer subjects for facilitation of Enhanced EBRT | 3 months
Intraprostatic lesion delineation capabilities of 11C-Choline in selected prostate cancer subjects for facilitation of Enhanced EBRT | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Amanie, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada